CLINICAL TRIAL: NCT00561743
Title: A Phase II Study to Assess the Safety and Efficacy of DBd Combination Therapy (DOXIL/CAELYX) [Doxorubicin HCL Liposome Injection], VELCADE [Bortezomib] and Dexamethasone) for Previously Untreated Multiple Myeloma Patients
Brief Title: A Study Assessing Safety and Effectiveness of BORTEZOMIB Combination Therapy (Bortezomib + Doxorubicin Hydrochloride + Dexamethasone) in Previously Untreated Multiple Myeloma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR010927
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2010-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; response rate; peripheral stem cell transplant; safety; tolerability
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone

INTERVENTIONS:
Drug: Bortezomib + pegylated liposomal doxorubicin HCl + dexamethasone

SUMMARY:
The purpose of this study is to determine whether doxorubicin HCL liposome injection, bortezomib, and Dexamethasone in combination, are effective in previously untreated multiple myeloma patients. Bortezomib inhibits the function of proteasomes, a novel mechanism of action.

DETAILED DESCRIPTION:
This was a single-arm, open-label, Phase II multi-centre study in Canada only. A total of 50 newly diagnosed multiple myeloma patients who were eligible for stem cell transplant were targeted for recruitment to this study. Combination doxorubicin HCL liposome injection, bortezomib and dexamethasone induction therapy was given for 4 cycles in preparation for stem cell collection and transplant. As remission status after induction and prior to the first or second auto-transplant has been shown to be the major determinant of both event free and overall survival in multiple myeloma patients, the goal has been to improve response rates through the use of various combinational approaches. As such, the objective of the present study was to test the hypothesis that treatment with this regimen could result in a higher complete + near complete response rate (CR + nCR) prior to stem cell transplant, than obtained with current regimens, and then to confirm the response rate post-transplant. Safety was evaluated using adverse event reportings, clinical laboratory tests and tests for cardiac function (multiple-gated acquisition scan/echocardiogram and electrocardiogram). Four 21-day cycles of combination induction therapy consisting of 1.3 mg/m2 bortezomib (given i.v. Days 1, 4, 8, 11) + 30 mg/m2 Doxil/Caelyx (given i.v. Day 4) + 40 mg Dex (given po Days 1-4, 8-11, 15-18 Cycle 1 only; Days 1-4 Cycles 2-4).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with newly diagnosed multiple myeloma (MM) requiring therapy for whom stem cell transplantation is considered appropriate
* Normal left ventricular ejection fraction
* Able to give voluntary written informed consent
* Female patients agree to use acceptable method for contraception

Exclusion Criteria:

* Diagnosis of smoldering multiple myeloma (asymptomatic MM with absence of lytic bone lesions)
* Renal insufficiency related to the monoclonal protein
* Diagnosis of Waldenström's disease
* Previous treatment for MM (excepting emergency use of a short course dexamethasone, radiation received > 30 days before study enrolment, plasmapheresis for treatment of clinically significant hyperviscosity syndrome > 30 days before trial enrolment)
* Major surgery within 30 days before entry
* Peripheral neuropathy or neuropathic pain Grade 2 or higher within 14 days of trial enrolment
* Uncontrolled or severe cardiovascular disease (including myocardial infarction within 6 months prior to enrollment
* NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, cardiac amyloidosis, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities)
* Other malignancy within the past 5 years prior to enrolment (except for non-active basal cell or non-metastatic squamous cell carcinoma of the skin, cervical carcinoma in situ or Stage 1 carcinoma of the cervix
* Known HIV seropositivity or active hepatitis A, B, or C infection
* Use of any investigational drug within 30 days prior to enrolment in the trial
* Medical or psychiatric condition that could interfere with trial participation
* History of hypersensitivity or allergic reaction attributable to compounds containing boron, mannitol or doxorubicin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was complete response (CR) and near complete response rate (nCR) post induction therapy (i.e. 4 cycles of therapy). Each cycle consisted of 21 days.

SECONDARY OUTCOMES:
The secondary endpoints included time to best response, assessment of peripheral blood stem cells harvesting ( 3 weeks post cycle 4 day 21) and engraftment (within 4 weeks of mobilization), CR post-engraftment, QoL and safety (every cycle).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada